CLINICAL TRIAL: NCT03742609
Title: A Randomised Controlled Trial of a Self-management Intervention for Adult Patients With Hearing Difficulties to Promote Hearing Aid Use and Benefit.
Brief Title: A Self-management Intervention for Adult Patients With Hearing Difficulties to Promote Hearing Aid Use and Benefit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Noor Afzarini Hasnita Binti Ismail, Principle Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 234737
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Written Information; Written Info and Hearing Aid Reminder; Written Info and Planning on Hearing Aid Use; All Materials

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Information only (No Intervention): provision of written information regarding consequences of using a hearing aid and not using a hearing. For example using a hearing aid will improve ability to hear others.
- Physical reminder only (Active Comparator): provision of written information regarding consequences of using a hearing aid and not using a hearing and physical reminder to use a hearing aid. For example, a hearing aid box as a physical reminder to use the hearing aids.
  Interventions: Other: ii) the reminder
- Behaviour Plan only (Active Comparator): provision of written information regarding consequences of using a hearing aid and not using a hearing and creation of behaviour plan to use a hearing aid. For example, when and where to use the hearing aids.
  Interventions: Other: ii) written behavioural plan
- Info, Reminder and Plan (Experimental): provision of written information regarding consequences of using a hearing aid and not using a hearing, physical reminder and creation of behaviour plan to use a hearing aid
  Interventions: Other: iv) all materials

INTERVENTIONS:
Other: ii) the reminder — Participants assigned to the prompt group were received instruction to use their hearing aid box as a physical prompt to remind participants to use their hearing aid(s)
  Arms: Physical reminder only
Other: ii) written behavioural plan — Participants assigned to this group were received instruction to create at least one written plan for hearing aid use. Specifically, participants were asked to plan where and when to use their hearing aid(s).
  Arms: Behaviour Plan only
Other: iv) all materials — i) provision of written information regarding consequences of using a hearing aid and not using a hearing aid, ii) the provision of a physical prompt for the purpose of prompting or cueing the behavior (hearing aid use) development, and iii) creation of a written behavioural plan for hearing aid use.
  Arms: Info, Reminder and Plan

SUMMARY:
The aim of the present study is to test I-PLAN as a self-management tool to promote hearing aid use and benefit (measured by self-reported questionnaires and hearing aid data-logging) among new adult hearing aid patients via a randomised controlled trial compared to treatment as usual. We hypothesized that the I-PLAN will increase hearing aid use and reduce self-reported hearing difficulty via promoting hearing aid use habits and self-regulation with respect to hearing aid use.

DETAILED DESCRIPTION:
The aim of the present study is to test I-PLAN, an intervention designed to promote hearing aid use among adult hearing aid patients, for the first time. I-PLAN is the first intervention in audiology that has been developed using the behaviour change wheel. It consists of three components; i) provision of written information regarding consequences of using a hearing aid and not using a hearing aid, ii) the provision of a physical prompt for the purpose of prompting or cueing the behavior (hearing aid use) development, and iii) creation of a written behavioural plan for hearing aid use.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or above
2. Have never used a hearing aid before
3. Have good understanding of English
4. have sufficient mental capacity to provide informal consent based on audiologist's opinion

Exclusion Criteria:

1. Have inability to complete the questionnaires due to age-related problems (for example; dementia) based on audiologist's opinion
2. presence of medical contraindications for hearing aids as described by the British Academy of Audiology (BAA, 2007)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Hearing aid use | 6-weeks
  Self-reported hearing aid use

CONTACTS AND LOCATIONS:
Overall Officials: Piers Dawes, Dr, Principal Investigator — Manchester Centre for Audiology and Deafness,University of Manchester
Locations (1):
- Audiology Clinic, Manchester, United Kingdom

REFERENCES:
- [Derived] Ismail AH, Armitage CJ, Munro KJ, Marsden A, Dawes PD. Evaluation of the I-PLAN Intervention to Promote Hearing Aid Use in New Adult Users: a Randomized Controlled Trial. Ear Hear. 2022 Jul-Aug 01;43(4):1103-1113. doi: 10.1097/AUD.0000000000001195. Epub 2022 Jan 6. PMID 34999593